CLINICAL TRIAL: NCT03777280
Title: Evaluation of Retention of Partial Denture Made of Injection Molded PEEK Framework Versus Cobalt Chromium Framework in Mandibular Kennedy Class I Edentulous Cases
Brief Title: Comparison Between Injection Molded PEEK Framework and Cobalt Chromium Framework in Removable Partial Denture Regarding Retention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haytham Mohammed talaat ahmed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-11-27
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Mandibular Prosthesis User

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peek framework Removable partial denture (Experimental): polymer-based framework has recently been introduced which is made of polyetheretherketone polymer frame combined with acrylic resin denture teeth and a conventional acrylic resin denture base.
  Interventions: Device: peek framework RPD
- cobalt chromium framework Removable partial denture (Active Comparator): it's the gold standard framework which has many benefits such as they are used in thin sections and are less bulky,provide high strength and stiffness,and some disadvantages include hypersensitivity,metal display and oral galvanism,
  Interventions: Device: cobalt chromium framework RPD

INTERVENTIONS:
Device: peek framework RPD — it is a polyetheretherketone polymer frame combined with acrylic resin denture teeth and a conventional acrylic resin denture base made by injecting technique and have several advantages regarding strength and esthetics
  Arms: peek framework Removable partial denture
Device: cobalt chromium framework RPD — standard framework device
  Arms: cobalt chromium framework Removable partial denture

SUMMARY:
This study is aiming to evaluate the retentive forces in PEEK framework RPD compared to Cobalt-Chrome framework RPD during attachment/detachment cycles in mandibular kennedy class I edentulous cases

ELIGIBILITY:
Inclusion Criteria:

* . kennedy class I edentulous subjects indicated for framework partial denture

Exclusion Criteria:

* Uncooperative patients and bad oral hygiene patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Retention | change from baseline retention force after one month and after three months
  retention force of RPD during attachment/detachment cycles measured by digital force meter device

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Souza JE, Silva NR, Coelho PG, Zavanelli AC, Ferracioli RC, Zavanelli RA. Retention strength of cobalt-chromium vs nickel-chromium titanium vs CP titanium in a cast framework association of removable partial overdenture. J Contemp Dent Pract. 2011 May 1;12(3):179-86. doi: 10.5005/jp-journals-10024-1031. PMID 22186813